CLINICAL TRIAL: NCT03622723
Title: Does the Radiological Stage Allow to Predict the Efficacy of an Intra-articular Injection of Hyaluronic Acid Among Patients Affected by a Hallux Rigidus ?
Brief Title: Radiological Stage and Efficacy of an Intra-articular Injection of Hyaluronic Acid for the Treatment of Hallux Rigidus
Acronym: REPAR
Status: Completed | Type: Observational
Sponsor: Labrha (Industry)
Responsible Party: Sponsor
Other Study IDs: 2015-A01904-45
Record Dates: First submitted 2018-03-05; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Hallux Rigidus, Unspecified Foot
Keywords: hallux rigidus; viscosupplementation; hyaluronic acid; metartarsophalangeal joint; foot arthritis; osteoarthritis of the big toe
MeSH Terms: conditions — Hallux Rigidus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The hallux rigidus is the most frequent type of arthrosis at the age of 50 and beyond. For the moderate forms of the disease, the majority of the studies recommend the recourse to the viscosupplement because of its efficiency in the long term.

On the other hand, no study was focused on the impact of the anatomical severity on the clinical result of the treatment by intra-articular injection of hyaluronic acid.

The present research has for objective to study the influence of the radiological severity on the result of the viscosupplement, in the conditions of daily practice, in patients affected by Hallux rigidus.

It is an open observational multicentrical prospective study realized by 20 investigators rheumatologists and liberal orthopedic surgeons. The recruitment is competitive and the study will be ended when 66 patients will have been included by taking into account a risk of trial exits or of lost of sight of 10 %.The main criterion is the influence of the radiological stage on the answer to the treatment.

Duration of inclusion 6 months. Duration of follow-up 3 months. Total duration of the study 9 months.

DETAILED DESCRIPTION:
Sixty patients presenting a hallux rigidus asserted by radiography and justifying a viscosupplement, without other selection criterion than the opinion of the investigator concerning the legitimacy of a viscosupplement and the agreement of the patient participating in the study.

The data collected during the consultations at J0 and J90 will be inputed by the investigator in the paper version of the CRF.

The informations collected during the initial consultation (J0) are: demographic (sex, age, weight, size), pathological (history of the disease, bilaterality, surgery of the big toe, evaluation of pain at J0 (scale of Likert : 11 points), treatments with analgesic aim, use of an orthosis), radiologics (Dell's stage), techniques (type of radiological or ultrasound guide).

The informations collected during the final consultation (J90) are: the evaluation of pain at J90 (scale of Likert 11 points), the perception by the patient of the efficiency of the treatment at J90 (scale of Likert 4 points), variation of its consumption of analgesic or of AINS (scale of Likert 3 points).

A descriptive analysis will be performed to characterize the demographic data, the history of the disease and its treatments, as well as the clinical and radiological data of the patients in the date of the inclusion.

The answer to the treatment will be estimated by 2 modalities (YES/NO) from the answer of the patients at the question " How do you judge the efficiency of the treatment ?": yes if the patients answered "Effective" or "very effective", no if they answered "little effective" or "not effective".

The influence of the radiological stage on the answer to the treatment will be studied (main criterion). The influence of radiological stage on the level of pain at J0 and on the reduction of pain between J0 and J90 will also be studied.

The coefficients of the multivariate models (ANCOVA and mixed model) will be considered as significant if their p-value is inferior to the threshold of 5%.

ELIGIBILITY:
Inclusion Criteria:

* • Patients of both genders, of all ages

  * Hallux rigidus confirmed by radiography including frontal and side radiographies performed during the last 6 months
  * Patients requiring a viscosupplement based on the opinion of the investigator
  * Patients were able to read and understand the information sheet, to give their enlighted consent and to respect follow up consultations

Exclusion Criteria:

* Patient with hypersensitivity to hyaluronic acid or mannitol
* Patient with a contraindication to the injection procedure : infected skin lesions on or close to an injection site, infectious disease ongoing
* Patient who received a viscosuplement during the last 3 months
* Patient who received an intra-articular injection of corticoids in the target articulation during the month before the inclusion
* Patient not talking french
* Patients that must undergo a surgical operation planned during 3 months following the injection susceptible to interfere with the follow-up or the evaluation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sixty patients presenting a hallux rigidus asserted radiologically and justifying according to the opinion of the rhumalologist or the surgeon a viscosupplementation. The study is realized in the conditions of daily practice, it modifies not at all the therapeutic care of the patient
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2016-04-19; Primary Completion 2018-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Correlation between the radiological stage and the treatment response | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: thierry CONROZIER, MD, Principal Investigator — Labrha
Locations (1):
- LABRHA, Lyon, France

IPD SHARING:
Plan to Share IPD: No